CLINICAL TRIAL: NCT04603053
Title: Acceptability and Effectiveness of an mHealth Intervention to Provide Cognitive Behavioral Therapy (CBT) for Adolescents With Depression/Anxiety
Brief Title: Determining Effectiveness of an mHealth Intervention to Provide Adolescent CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Washington University Institute of Clinical and Translational Sciences (Unknown)
Responsible Party: Principal Investigator, Jane Garbutt, MD, Professor of Medicine and Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202005103
Record Dates: First submitted 2020-10-16; First posted 2020-10-26 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Adolescent Depression; Anxiety Disorders
Keywords: Cognitive Behavioral Therapy; mHealth
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBot-A Group (Experimental): Participants randomly assigned to this arm will receive access to CBot-A app.
  Interventions: Behavioral: mHealth app
- Wait List Group (No Intervention): Participants randomly assigned to this arm will be offered the intervention after the completion of the trial.

INTERVENTIONS:
Behavioral: mHealth app — Participants will receive access to CBot-A app for 12 weeks.
  Arms: CBot-A Group

SUMMARY:
Washington University will evaluate the acceptability and effectiveness of a mobile health (mHealth) intervention to provide cognitive behavioral therapy for adolescents with depression.

DETAILED DESCRIPTION:
In this pilot project, Washington University will start to evaluate CBot-A, a promising mHealth therapeutic intervention designed to deliver cognitive behavioral therapy (CBT) through an app on a phone or other mobile device. The evaluation will include a randomized trial among 40 adolescents diagnosed with depression and/or anxiety and will assess if CBot-A is usable by teens and likely to provide benefit, and acceptable to adolescents.

The primary outcome of depression and anxiety symptoms in adolescents will be assessed at 1 month and 3 months to check for any changes.

ELIGIBILITY:
Inclusion Criteria:

Adolescents 12-17 years of age and diagnosed with a major depressive disorder (MDD) and/or generalized anxiety disorder by their primary care provider within the past 3 months.

Exclusion Criteria:

Adolescents with the following conditions (identified by parental report) will be excluded:

* Participated in formal CBT within the past 12-months
* Diagnosed with severe depression
* Diagnosed with the following anxiety disorders - obsessive-compulsive disorders, post-traumatic stress disorder, panic disorder, or specific phobias
* A psychiatric hospitalization in the previous month
* With significant comorbidities such that the PCP would refer to a mental health professional for treatment, including those with a substance use disorder or a psychotic illness.
* Are not accompanied by a guardian to the diagnostic visit
* Without access to a mobile device (cell phone or tablet) for regular use
* Unable to read and write English
* Participants may also be excluded at the discretion of the PI.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 1 month
  The PHQ-9 Adolescent Version will be used.This 9-item instrument scores from 0 to 27, with higher scores indicating more depressive symptoms

SECONDARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) | 1 month
  This 7 item instrument scores from 0 to 21 with higher scores indicating more anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jane Garbutt, MB, ChB, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Nicol G, Wang R, Graham S, Dodd S, Garbutt J. Chatbot-Delivered Cognitive Behavioral Therapy in Adolescents With Depression and Anxiety During the COVID-19 Pandemic: Feasibility and Acceptability Study. JMIR Form Res. 2022 Nov 22;6(11):e40242. doi: 10.2196/40242. PMID 36413390